CLINICAL TRIAL: NCT02016833
Title: Phase 0 Study for the Development of Immunological Assays for the Evaluation of WT-1, Survivin and HPV16 E7 Tumor Antigens Specific Immune Responses in Cancer Patients
Brief Title: Development of Immunological Assays for the Evaluation of Tumor Antigen Specific Immunity
Status: Completed | Type: Observational
Sponsor: PX Biosolutions (Industry)
Responsible Party: Sponsor
Other Study IDs: PX_DCtagTM_LeadIn_001
Record Dates: First submitted 2013-12-05; First posted 2013-12-20 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Serous Adenocarcinoma; Undifferentiated Carcinoma of Ovary; Cervical Cancer; Cervical Intraepithelial Neoplasia, Grade 3; Acute Myeloid Leukemia; Chronic Myeloid Leukemia
Keywords: Ovarian Cancer; Cervical Cancer; Leukemia; Immunity; WT-1; Survivin; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Ovarian Neoplasms; Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — PBMCs isolated from whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer patients: Patient with histologically confirmed diagnosis of cervical cancer or cervical intraepithelial neoplasia (grade 3) or of high-grade serous (or undifferentiated) ovarian cancer or patients with AML or CML confirmed by bone marrow biopsy or peripheral blood Not treated - prior standard of care therapy acceptable one blood sampling performed on the visit day
  Interventions: Procedure: Blood Sampling

INTERVENTIONS:
Procedure: Blood Sampling — Sampling of 80mL of whole blood

SUMMARY:
This study is a clinical study aiming at establishing immunological assays for the qualitative and quantitative evaluation of WT-1, Survivin and HPV16 E7-specific immune responses in cancer patients. Such a study will allow the development of suitable immunological tools to be used in assessing response in a subsequent phase I study aiming at evaluating therapeutic vaccine candidates targeting WT-1, Survivin and/or HPV16 E7-expressing tumors. In addition, this study will help defining the baseline cancer-associated immune responses in the selected patient population.

Cervical and ovarian cancer patients, as well as leukemia patients, will be included in this study.

WT-1, Survivin and HPV-specific immune responses will be monitored in these patients by ex vivo and cultured IFNg ELISpot as well as tetramer staining.

ELIGIBILITY:
Inclusion Criteria:

* Specific Inclusion criteria
* For ovarian cancer patients: Histologically confirmed surgical diagnosis of high-grade serous (or undifferentiated) ovarian cancer
* For CIN3 and cervical cancer patients: Histologically confirmed diagnosis of CIN3 or cervical cancer
* For AML and CML patients: HLA-A2 positivity and diagnosis of AML or CML confirmed by bone marrow biopsy or peripheral blood
* Shared inclusion criteria
* No evidence of active progressive disease. For ovarian cancer patients, a woman with a rising CA125 and negative imaging is acceptable
* Age ≥ 18 yrs and < 70 yrs
* ECOG 0-2
* Adequate hematologic assessment (results from the previous standard of care visit):
* Absolute neutrophil count (ANC) greater than or equal to 1.0 x 109/L
* Platelets greater than or equal to 100 x 109/L.
* Written informed consent

Exclusion Criteria:

* Treatment with chemotherapy, radiation therapy, other immunotherapy or non-topical steroids within the past 3 weeks prior to initiation of the study.
* Immunosuppressive therapy (excluding topical steroids) for any other condition.
* Recurrent/progressive disease confirmed clinically, radiologically or histologically before entry into the study. (exclude versus inclusion criteria)
* Persistent fever (>24 hours) documented by repeated measurement or active uncontrolled infection in the last 4 weeks.
* Active autoimmune disease, including, but not limited to, SLE, MS, ankylosing spondylitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three type of patients will be enrolled in this study:
  * Women with a confirmed diagnosis of serous or undifferentiated ovarian cancer
  * Women with a confirmed diagnosis of CIN3 or cervical cancer
  * HLA-A2 positive men or women with a confirmed diagnosis of AML of CML All these patients will be less than 70 years of age and will show no evidence of active progressive disease on follow up. For ovarian cancer patients, a woman with a rising CA125 and negative imaging is acceptable.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Development and validation of ELISpot and tetramer assays for the detection of tumor-antigen specific T cell immune responses in cancer patients | Baseline
  Direct and cultured IFNg ELISpot as well as direct tetramer staining assays will be set up and qualified for the detection WT-1, survivin and HPV16 E7 specific immune responses in cancer patients

SECONDARY OUTCOMES:
Characterisation of WT1, Survivin and HPV16 E7 specific immune responses in cancer patients | Baseline
  Direct and Cultured IFNg ELISpot assays as well as tetramer staining assays will be used for the characterization of tumor specific immune responses in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Linda Mileshkin, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Center, Melbourne, Victoria, Australia